CLINICAL TRIAL: NCT04270487
Title: A Randomized Controlled Trial to Evaluate the Short-term Efficacy and Long-term Health Economic Impact of a Dietary Intervention Compared to Pharmacotherapy With a Musculotropic Spasmolytic Agent for Newly Diagnosed or Newly Treated Irritable Bowel Syndrome in Primary Care
Brief Title: The DOMINO Trial: Diet Or Medication in Irritable Bowel syNdrOme
Acronym: DOMINO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S59482
Record Dates: First submitted 2019-09-27; First posted 2020-02-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — octylonium

STUDY DESIGN:
Intervention Model Description: Randomized Parallel study: diet vs medication (otilonium bromide)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS diet (Experimental): The simple IBS diet is a diet based on the Low FODMAPs diet and the NICE (National Institute of Health and Care Excellence) IBS diet. Patients will be aid to follow the diet with a mobile app.
  Interventions: Other: IBS Diet
- Otilonium bromide (Active Comparator): Otilonium bromide is a a frequently used musculotropic spasmolytic. The dosis used will be 40 mg t.i.d.
  Interventions: Drug: Otilonium Bromide

INTERVENTIONS:
Other: IBS Diet — Patients will be randomized to a diet or a mediation treatment
  Arms: IBS diet
Drug: Otilonium Bromide — Patients will be randomized to a diet or a mediation treatment
  Arms: Otilonium bromide

SUMMARY:
A randomized controlled trial to evaluate the short-term efficacy and long-term health economic impact of a dietary intervention compared to pharmacotherapy with a musculotropic spasmolytic agent for newly diagnosed or newly treated irritable bowel syndrome in primary care.

DETAILED DESCRIPTION:
A randomized controlled trial (Phase IV trial) to evaluate the short-term efficacy and long-term health economic impact of a dietary intervention compared to pharmacotherapy with a musculotropic spasmolytic (otilonium bromide) agent for 470 newly diagnosed or newly treated irritable bowel syndrome patients in primary care.

The primary objective of this trial is to study treatment efficacy (IBS-SSS responder rate) with diet versus medication after 8 weeks of therapy.

The secondary endpoint is to study the quality of life and health economic impact over six months after the start of the initial treatment with diet versus medication.

Finally, patient satisfaction during and after the different treatment modalities, HRU and WPAI-IBS score in subgroups according to IBS stool pattern subtype, faecal microbiota and serotonin synthesis genetic polymorphisms will also be investigated

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those of either gender, above the age of 18, eligible to give informed consent.
* Newly diagnosed with or newly to be treated for IBS in primary care, as this is the setting where the majority of these patients is managed. The diagnostic gold standard, in line with clinical practice, will be clinician's diagnostic judgment.
* Supportive information for the diagnosis of IBS will be provided to the GPs at the initial investigators meeting. This includes: a guidance for diagnosis and potentially useful additional tests based on the Rome IV management algorithm, a Rome IV-based diagnostic questionnaire with pictograms and a list of alarm symptoms.
* Patients who did not receive treatment over the preceding 3 months, and who did not receive long-term treatment (>3 consecutive weeks) with otilonium bromide in the past are eligible for the trial.

Exclusion Criteria:

* Patients not capable to understand or be compliant with the study.
* Patients with concurrent organic gastrointestinal disease (inflammatory bowel disease), a history of major bowel surgery (not including minimal invasive surgery such as appendectomy or cholecystectomy, but including sigmoidectomy, hemicolectomy and small bowel resections)
* Patients who received treatment with otilonium bromide in the past for more than 3 weeks consecutively or who received otilonium bromide recently for any duration in the last 3 months.
* Patients who have used FODMAP or NICE diet before.
* Patients who recently (last 3 weeks) used other medication for IBS, or who changed their diet for IBS or for any other reason over the last 3 months. To be included in the trial patients should stop these treatments following the advice of their GP (see paragraph 8.9).
* Patients with diabetes, uncontrolled thyroid disease, active malignant disease (not including patients with cancer free diagnosis for more than 5 years), symptomatic uncontrolled endometriosis.
* Patients with a major psychiatric disease. The use of a single antidepressant on a stable dose for at least 3 months is allowed (see paragraph 8.9).
* Patients with drug abuse and/or alcohol abuse.
* Patients on pharmacologically prepared probiotic formulations (i.e. bought in the pharmacy) will be excluded. The use of probiotic drinks or yoghurts available from food stores, such as Activia®, Yakult ®, Actimel ®, is allowed but should be registered as "complementary treatment"(see paragraph 8.9).
* Women with active pregnancy plans in the coming 6 months are not eligible and women of childbearing potential are only eligible if they use effective contraception throughout the study. Also excluded are women of childbearing potential not using effective contraception or women planning to become pregnant the next 6 months (see paragraph 8.9). Methods of contraception considered highly effective are: combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, a vasectomized partner or sexual abstinence (http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy of symptom severity | 1.5 year
  IBS-SSS: IBS symptom severity score
  The maximum achievable score is 500. Mild, moderate and severe cases were indicated by scores of 75 to 175, 175 to 300 and >300 respectively.
  Controls scored below 75 and patients scoring in this range can be considered to be in remission.
  Efficacy of treatment will be assess by calculating the proportion of patients in each arm with a drop of 50 points or more on the IBS-SSS. The higher the drop, the more the patient has improved.

SECONDARY OUTCOMES:
Treatment efficacy in quality of life | 1.5 year
  Assessment will be done with the IBS-QoL questionnaires before and during the study.
  This includes IBS generic functional status and well-being, perceived quality of life specific to IBS, and work disability.
  Quality of life and health economic impact over 6 months after the start of the initial treatment with diet versus medication will be studied.
  Questionnaire includes a 5-point Likert response scale: not at all, slightly, moderately, quite a bit, and extremely or a great deal.
  All items were sum-scored to calculate total scores.

OTHER OUTCOMES:
Quality of life in IBS | 1.5 year
  Euro-Qol quesrionnaire. This questionnaire includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 3 levels: no problems, some problems, extreme problems.
  Additionallty, a VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
  All the scores are taken into account.
Work Productivity and Activity Impairment in IBS | 1.5 year
  Work Productivity and Activity Impairment Questionnaire (WPAI) Levels of work productivity will be assess before and after treatment. The change of work productivity levels before and after treatment will be studied.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Questions:
  1. = currently employed
  2. = hours missed due to health problems
  3. = hours missed other reasons
  4. = hours actually worked
  5. = degree health affected productivity while working
  6. = degree health affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages. Percent work time missed due to health: Q2/(Q2+Q4) Percent impairment while working due to health: Q5/10 Percent overall work impairment due to health: Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)] Percent activity impairment due to health: Q6/10
Depression levels in IBS | 1.5 year
  PHQ: patient health questionnaire
  This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of -not at all,‖ -several days,‖ -more than half the days,‖ and -nearly every day,‖ respectively.
  PHQ-9 total score (sum) for the nine items ranges from 0 to 27.
  Scores represent: 0-5 = mild 6-10 = moderate 11-15 = moderately severe 16-20 = severe depression
  Levels of depression will be assess before and after treatment. The change of depression levels before and after treatment will be studied.
Somatic levels in IBS | 1.5
  PHQ: patient health questionnaire
  This is calculated by assigning scores of 0, 1, and 2 to the response categories of -not at all‖, -bothered a little‖, and -bothered a lot‖, for the 13 somatic symptoms and 2 items from the depression module (sleep and tired) are scored 0 (-not at all‖), 1 (-several days‖) or 2 (-more than half the days‖ or -nearly every day‖).
  PHQ-15 scores (sum of scores) of 5, 10, and 15 represent cutpoints for low, medium, and high somatic symptom severity, respectively.
  Levels of somatization will be assess before and after treatment. The change of somatization levels before and after treatment will be studied.
Anxiety levels in IBS | 1.5 years
  GAD-7 - patient health questionnaire This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively. GAD-7 total score for the seven items ranges from 0 to 21. When screening for anxiety disorders, a recommended cutpoint for further evaluation is a score of 10 or greater.
Health resourse utilisation in IBS | 1.5 years
  Health resourse utilisation in IBS with the HRU questionnaire. Both direct and indirect health costs, including self-costs to patients, will be compared at the different time points (2,4,6 months). They will also be compared to the (retrospective) cost assessment at baseline. The total direct costs of the utilization of healthcare resources associated with IBS will be calculated in terms of (additional) primary care visits, secondary care visits, hospitalizations, diagnostic tests and procedures, prescription and non-prescription medication and complementary therapies.
Genetic prediction to treatment in IBS | 1.5 years
  Exploratory outcome GWAS analysis of IBS genetics. Pathophysiological and treatment predictors will be investigated in an exploratory setting
Microbiome prediction to treatment in IBS | 1.5 years
  Exploratory outcome Microbiome analysis of IBS stool samples. Pathophysiological and treatment predictors will be investigated in an exploratory setting

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Univeristy Hospital Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Tack C, Van den Houte K, Besard L, Capiau L, Ceulemans S, Gernay O, Maes S, Peetermans C, Raat W, Stubbe J, Van Boxstael R, Vandeput O, Van Steenbergen S, Gehesquiere B, Raes J, Tack J, Carbone F. A study on the utility of inflammatory biomarkers in primary care irritable bowel syndrome: a sub analysis of the DOMINO randomized trial. BMC Gastroenterol. 2025 Dec 23. doi: 10.1186/s12876-025-04494-7. Online ahead of print. PMID 41436948
- [Derived] Di Rosa C, Van den Houte K, Altomare A, Guarino MPL, Besard L, Arts J, Caenepeel P, Piessevaux H, Vandenberghe A, Matthys C, Biesiekierski JR, Capiau L, Ceulemans S, Gernay O, Jones L, Maes S, Peetermans C, Raat W, Stubbe J, Van Boxstael R, Vandeput O, Van Steenbergen S, Van Oudenhove L, Vanuytsel T, Jones M, Tack J, Carbone F. DOMINO trial post hoc analysis: evaluation of the diet effects on symptoms in IBS subtypes. Therap Adv Gastroenterol. 2024 Jul 30;17:17562848241255296. doi: 10.1177/17562848241255296. eCollection 2024. PMID 39086991
- [Derived] Carbone F, Van den Houte K, Besard L, Tack C, Arts J, Caenepeel P, Piessevaux H, Vandenberghe A, Matthys C, Biesiekierski J, Capiau L, Ceulemans S, Gernay O, Jones L, Maes S, Peetermans C, Raat W, Stubbe J, Van Boxstael R, Vandeput O, Van Steenbergen S, Van Oudenhove L, Vanuytsel T, Jones M, Tack J; DOMINO Study Collaborators; Domino Study Collaborators. Diet or medication in primary care patients with IBS: the DOMINO study - a randomised trial supported by the Belgian Health Care Knowledge Centre (KCE Trials Programme) and the Rome Foundation Research Institute. Gut. 2022 Nov;71(11):2226-2232. doi: 10.1136/gutjnl-2021-325821. Epub 2022 Apr 28. PMID 35483886